CLINICAL TRIAL: NCT01910844
Title: Phase II Pilot Study Assessing Efficacy of a Cisplatin - Métronomic Cyclophosphamide Treatment in Patients With Stade IV Triple Negative Breast Cancer Secondary Resistant to Anthracyclines and Taxanes
Acronym: META2
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Because of difficulties in recruting
Sponsor: Centre Jean Perrin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CJP 4.2 - META2
Record Dates: First submitted 2013-05-28; First posted 2013-07-30 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-07

CONDITIONS: Metastatic Breast Cancer
Keywords: triple negative breast cancer; late-relapse
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Cisplatin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cisplatin - Metronomic Cyclophosphamide (Experimental): Cisplatin 25 mg/m² from day 1 to day 3 every 3 weeks Metronomic Cyclophosphamide 150 mg from day 1 to day 14 every 3 weeks
  Interventions: Drug: Cisplatin; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Cisplatin — 25 mg/m² I.V. from day 1 to day 3 - total dose = 75 mg/m² every 3 weeks
Drug: Cyclophosphamide — Metronomic cyclophosphamide per os 150 mg from day 1 to day 14 - total dose 2100 mg every 3 weeks
  Other Names: Endoxan

SUMMARY:
Study assessing efficacy of a Cisplatine- Métronomic cyclophosphamide treatment in Patients with Metastatic Triple Negative breast Cancer Secondary Resistant to Anthracyclines and Taxanes.

ELIGIBILITY:
Inclusion Criteria:

* Performance status < 2,
* Patient with metastatic breast cancer stade IV triple negative histologically confirmed
* Measurable or not disease but radiologically evaluable (RECIST 1.1),
* Negative Hormonal Receptors (Estrogens and/or Progesterone),
* HER-2 negative (Score 0 or 1 by Immunochemistry (IHC), negative FISH if score IHC 2),
* Patient exposed to anthracyclines and/or taxanes in neo-adjuvant or adjuvant setting,
* Patient with a progression and for whom anthracyclines and/or taxanes treatment cannot be delivered and according to a resistance defined as :
* In the last 12 months after the last dose of taxanes or anthracyclines in adjuvant or neoadjuvant setting or,
* During or after a first metastatic chemtotherapy line and where taxanes and anthracyclines cannot be delivered according to :
* either a secondary resistance after an initial response to chemotherapy but a relapse observed either during the treatment or in the 4 months after the end of chemotherapy.
* either a sensitivity to treatment defined by a relapse after more than 4 months after the first chemotherapy metastatic line,
* either intolerance to anthracyclines (doxorubicin 240-400 mg/m² ou equivalent to doxorubicin (epirubicin) 300-550mg/m²)
* Patient non previously treated by platinum salts,
* Hematological Functions: Neutrophiles ≥ 1,5.109/L, Platelets ≥ 100.109/L, Leucocytes > 3 000/mm3, Hb > 9g/dL, Hepatic Functions : total Bilirubin ≤ 1,5 time upper normal value (UNV), ASAT ≤ 2 ,5 time UNV, ALAT ≤ 2,5 time UNV, Alkaline Phosphatase ≤ 2,5 time UNV (< 5 time UNV if case of hepatic metastasis), Renal Functions: Serum Creatinine ≤ 1,5 time UNV (and if value > 1,5 time UNV, so Clearance ≥ 60 mL/min) or Clearance ≥ 40 mL/min in case of RMI,
* Patient signed the consent study form,
* Patient affiliated to a social security regimen (law of 9 August 2004).

Exclusion Criteria:

* Male Patients,
* Unknown hormonal Receptors
* Positive HER-2 (Score 3 in IHC or positive FISH)
* Pregnant or breastfeeding patient, or in age of pregnancy or predicting to be pregnant in the 6 months after the end of treatment,
* Patient not using contraceptive treatment during the treatment or after the 6 months after the end of treatment,
* Patient is a ward,
* Patient suffering from a non compatible disease with the enrollment in the study,
* Cardiac, renal, medullar, respiratory or hepatic insufficiency, clinically significant cardiovascular disease (including myocardiac infarct, unstable angina, symptomatic congestive heart failure, uncontrolled cardiac arrhythmia) < 1 year before the study enrollment or randomisation,
* Patient with pulmonary lymphangitis or symptomatic pleural effusion (grade≥2), meningeal known carcinoma or symptoms of cerebromeningeal invasion, brain metastases unless treatment and stability for at least 4 weeks (no steroids or anti-convulsive).
* Uncontrolled diabetes,
* Psychiatric or neurological significant abnormality,
* Peripheric Neuropathy > grade 2,
* Antecedent of hypersensibility to one of study treatment or one of used excipients,
* Urinary tract infection or acute hemorrhagic cystitis in progress
* Concomitant treatment with a medicine containing phenytoin or medication received in the context of a trial, or participation in another therapeutic clinical trial within <30 days prior treatment with chemotherapy.
* Geographically unstable patient in the next 6 months or remaining distance to the treatment center making it difficult to follow in the study,
* Known history of abuse of narcotic or other drug or alcohol
* History of surgery within 28 days before the start of treatment,
* Patient unwilling or unable to comply with the requirements of the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-07; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Response rate of cisplatine - metronomic cyclophosphamide treatment | 12 months and 6 weeks

SECONDARY OUTCOMES:
Disease free progression | 3 years
Safety profile of cisplatin - metronomic cyclophosphamide association | 12 months and 6 weeks
  Number of Participants with Adverse Events
Overall survival | 5 years
Predictive factors to response and/or resistance treatment | 12 months and 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Jean Perrin, Clermont-Ferrand, France